CLINICAL TRIAL: NCT04603651
Title: Expanded Access Information for Physicians for Bamlanivimab (LY3819253) Emergency Investigational New Drug [EIND]
Brief Title: Expanded Access Program to Provide Bamlanivimab (LY3819253) for the Treatment of COVID-19
Status: No longer available | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AbCellera Biologics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18165; J2X-MC-Y001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-10-23; First posted 2020-10-27 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09-15

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Bamlanivimab — Administered intravenously (IV).
  Other Names: LY3819253; LY-CoV555

SUMMARY:
The treating physician/investigator contacts Lilly when, based on their medical opinion, a patient meets the criteria for inclusion in the expanded access program.

ELIGIBILITY:
Inclusion Criteria:

* Reside in a country where there are ongoing Lilly-sponsored clinical trials (currently this is only the United States)
* Present within 10 days of symptom onset
* Have severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) confirmed by reverse transcription polymerase chain reaction (RT-PCR) within the last three days
* Participants greater than or equal to (≥) 65 years of age OR
* Participants ≥ 12 years of age who weigh at least 40 kilograms AND have at least one of the following:

  * Cancer
  * Chronic kidney disease
  * Chronic obstructive pulmonary disease (COPD) or other chronic lung disease
  * Immunocompromised state (weakened immune system or on immunomodulatory medications)
  * Obesity (body mass index [BMI] of 35 or higher)
  * Serious heart conditions such as heart failure, coronary artery disease or cardiomyopathies
  * Sickle cell disease
  * Diabetes mellitus (Types 1 or 2)

Exclusion Criteria:

* Require hospitalization greater than (>) 24 hours or hospice care. Residents in long term care or skilled nursing facilities that meet the inclusion criteria and are not on mechanical ventilation will be considered
* Bamlanivimab should not be used in patients hospitalized with severe COVID-19 respiratory disease

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Contact Lilly at 1-800-LillyRx (1-800-545-5979), Study Director — Eli Lilly and Company

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343